CLINICAL TRIAL: NCT02554071
Title: Manitoba Pharmacist Initiated Smoking Cessation Pilot Project
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Govenment of Manitoba (Unknown); Canadian Foundation for Pharmacy (Unknown); Neighbourhood Pharmacy Association of Canada (Unknown)
Responsible Party: Principal Investigator, Dr. Shawn Bugden, Associate Professor, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H2013:459
Record Dates: First submitted 2015-09-16; First posted 2015-09-18 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pharmacist - Smoking Cessation Support' (Experimental): Active Comparator Arm Receive smoking assessment Initial Smoking Cessation Counselling Smoking Cessation Prescription/Non-Prescription Product as required Follow-up Counselling
  Interventions: Other: Pharmacist - Smoking Cessation Support

INTERVENTIONS:
Other: Pharmacist - Smoking Cessation Support — Intervention mirrors clinical practice with smoking cessation counselling -- patients receive smoking cessation product at no cost and pharmacists are paid flat fee for providing counselling

SUMMARY:
A single arm pilot study conducted to assess the feasibility of having Manitoba Pharmacists provide support (product and cognitive) to low-income (receiving social assistance) smokers wishing to quit smoking.

DETAILED DESCRIPTION:
SYNOPSIS - Manitoba Pharmacist Initiated Smoking Cessation Program Overview Background The Manitoba government supports the role of the pharmacist as an integral part of the primary health care team delivering quality care and service to Manitobans. The role of the Pharmacist is ever evolving and expanding to meet the needs of their clients including comprehensive medication therapy management and expanded preventative expert. Community pharmacists are one of the most accessible health care professionals and provide a wide range of clinical services in the neighborhoods, towns, and cities across this province.

As part of the Manitoba government's wellness initiative, the government is strategically committed towards reducing the use of tobacco through public policy. Smoking is one of the leading causes of death in Manitoba and the use of tobacco is responsible for more than 50% of lung, respiratory, and oral cancers and a substantial factor in cardiovascular disease. While decreases in smoking rates have been achieved in recent years, Manitoba continues to exceed the national average of 17.3%, ranking the province with the third highest smoking prevalence. Manitoba' current smoking rates warrant continued efforts to reduce smoking in youth and adults.

While many believe smoking to be lifestyle choice it is also known to be a changeable lifestyle behavior and a significant determinant of health. It is also known to be a serious addiction that is very difficult to overcome both physically and emotionally. As part of Manitoba's targeted approach to smoking cessation, a partnership has been forged to develop and implement the pilot program: Manitoba Pharmacist Initiated Smoking Cessation Program.

Methodology The role of the pharmacist can best be described as underutilized and often an under recognized resource in smoking cessation programs. For individuals who smoke, many find smoking cessation overwhelming and difficult without assistance, including smoking cessation drugs and ongoing support and counselling. Many pharmacists have received additional knowledge and training specifically for initiating and monitoring a smoking cessation for individual clients. The Manitoba Pharmacist Smoking Cessation Program will provide access for 100 clients to the vital components necessary to quit smoking. Lower socioeconomic status is associated with higher rates of smoking. The Manitoba Employment and Income Assistance program provides support for lower income individuals in Manitoba. This smoking cessation program is a controlled pilot study providing clients with the most appropriate smoking cessation drugs along with the benefit of one to one pharmacist support and counselling.

Smoking Cessation Program Objectives

The following are the program objectives:

* Establish a provincial pilot smoking cessation program
* Reduce the number of Manitobans who smoke
* Enhance utilization of the pharmacist in preventative health care delivery

Program Scope A. Target Population

* 100 Manitoba residents over the age of 18 who are Manitoba Employment and Income Assistance active program participants as of January 01, 2014
* Provide written consent to participate in a smoking cessation program
* Agree to participate in the counselling sessions and smoking cessation behavior readiness
* Agree to participate in an evaluative process and follow up study

B. Participation Provider (Pharmacy and pharmacist)

1. Pharmacy/Pharmacists - Up to fifteen pharmacies throughout Manitoba who employ pharmacists professionally trained in QUIT and/or Catalyst, have previous experience providing smoking cessation services to patients, who are willing and able to commit to pilot project timelines, and who receive pharmacy manager approval will be eligible to apply to participate in this program.
2. In December 2013, MPhA will distribute application forms to each pharmacy for their voluntary consideration for participation and response to the call for applications. Each application form consists of a letter of introduction to explain the program and application process, a pharmacist manager application form, and pharmacist application form(s). The MPhA is the provincial regulatory body for pharmacists and pharmacies in Manitoba and thus has access to all pharmacy contact information. MPhA has agreed to utilize their mailing list and distribution system to communicate with all pharmacies in the province to ensure that equal access to any pharmacy and pharmacist in the province is achieved.
3. The Steering Committee will establish a Pharmacy Selection Sub-Committee to confidentially review all application forms for completeness and to select suitable complete a random selection process of all complete and eligible applications.
4. Up to 15 pharmacies in Manitoba who meet the provider eligibility criteria will be selected by the Pharmacy Selection Sub-Committee. All applicants will receive an outcome letter from the Program Manager following the selection process.
5. Successful pharmacy applicants will receive an orientation training program in the first week of January 2014 to share and educate pilot project details, participant recruitment processes, program implementation processes, methodology to complete participant informed consent and program surveys, evaluation requirements, and professional pharmacy reimbursement processes, and participant product reimbursement options.

Client Participation

1. Eligible participants in the pilot project include and Manitoba adult who meets the criteria of the targeted population cohort, and who have identified as being ready to quit smoking, will be eligible for the program.
2. Pharmacists participating as providers in the smoking cessation pilot project will be responsible for identifying eligible adults within their patient population as eligible for program participation.
3. All pharmacists in Manitoba are PHIA compliant.
4. Pharmacist providers will share with each potential participant a program information sheet, informed consent form, and access to a pharmacy staff person (pharmacy assistant/technician) not related to the pilot project and Pilot Project Project Manager contact information for access to pilot project information and independent decision making for project participation.
5. Completion of the Informed Consent Form will be independently completed by the potential applicant.
6. Support from an assigned pharmacy staff member not related to the pilot project will be made available should the potential applicant request.
7. Potential applicants will be encouraged to consult with their primary health care provider.
8. Each project participant:
9. Be introduced to the smoking cessation program and if interested given the informed consent to review. They may also be provided with some general educational materials on smoking cessation ii. Once the participant has had sufficient time to review the consent and has had all questions answered, the pharmacy assistant/technician will obtain informed consent.

iii. After consent has been obtained the patient will be provided with some forms to complete to assess their current smoking patterns and readiness to quit. When the completed forms are returned an initial assessment interview will be booked with the pharmacist.

iv. During the initial assessment interview:

1. The pharmacist will assess the level of dependence from the completed Fagerstrom Tolerance Scale and assess the motivations for smoking from the Why Test.
2. Potential drug interactions between medications and smoking/smoking cessation will be assessed.
3. The participant will be introduced to the Smoking Cessation Form and asked to record the symptoms, triggers, cessation product use and side effects on a daily basis.
4. The participant will be provided with a variety of educational materials to help guide their individualized quit plan (How Do I Want to Quit?, Why Do I Want to Quit?, When Do I Want To Quit?)
5. The pharmacist will work with the participant to complete the Pre-Quit Planning form
6. Additional Educational materials may be provided as needed ( Count Down to Quit Date, Breaking the Cycle of Addiction Date, My Reasons to Quit Smoking, Enlisting Support) v. Quit Day Visit:

1. The pharmacist will work with the participant to complete the Quit Day Plan. 2. The participant will be provided with the Quit Diary to record smoking 3. Additional Educational materials will be provided as needed (Managing Withdrawal Symptoms, Minimizing Weight Gain, Dealing with the Urge to Smoke, Managing Slips and Relapse, List of Resources).

4. Ensure the participant has a copy of the Smoking Cessation Assessment From for future telephone follow-ups.

vi. Phone Follow-up - 1 Week Post Quit

1. The pharmacist will provide telephone follow-up and review what has worked well and any challenges with withdrawal they have experienced. The Quit Plan will be modified as needed.
2. They will complete the Smoking Cessation Assessment Form with the patient. vii. 1 Month Post Quit Visit

1. The pharmacist will meet with the participant and review what has worked well and any challenges with withdrawal they have experienced. The Quit Plan will be modified as needed.

2. They will complete the Smoking Cessation Assessment Form with the patient. viii. 3 Month Quit Visit

1. The pharmacist will meet with the participant and review what has worked well and any challenges with withdrawal they have experienced. The Quit Plan will be modified as needed.
2. They will complete the Smoking Cessation Assessment Form with the patient.
3. Ensure the participant has a copy of the Smoking Cessation Assessment From for future telephone follow-ups.

ix. Phone Follow-up - 6 Month Post Quit

1. The pharmacist will provide telephone follow-up and review what has worked well and any challenges with withdrawal they have experienced. The Quit Plan will be modified as needed.
2. They will complete the Smoking Cessation Assessment Form with the patient.
3. Make a transition plan to ensure the participant has access to remaining to necessary support and suitable covered medications to maintain smoking cessation.

C. Program Duration Total duration of the study will be a 6-15 months. The participant will have access to smoking cessation pharmacy counseling services and smoking cessation products for a period of three months from the initiation in the pilot project. The intervention component of the pilot project will be available between January and April 2015.

ELIGIBILITY:
Inclusion Criteria:

* smoker
* >= 18 years
* receiving Manitoba Employment and Income Assistance as of January 1st 2015
* Stated desire to quit smoking
* Signed Consent with associated agreement to participate in evaluation and follow-up

Exclusion Criteria:

* < 18
* Not on Income Assistance
* Current non-smoker

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2014-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Smoking Cessation Assessment | 6 months
  Self-reported Smoking Cessation on Standardized Form

SECONDARY OUTCOMES:
Smoking Cessation Assessment | 1 month
  Self-reported Smoking Cessation on Standardized Form
Smoking Cessation Assessment | 3 months
  Self-reported Smoking Cessation on Standardized Form
Smoking Cessation Product | 3 months
  Smoking Cessation Product Used and Cost
Quit Diary | 6 months
  Record of Continued Smoking and Symptoms

OTHER OUTCOMES:
Cigarettes Smoked | day 0, 1 month, 3 months and 6 months
  # of cigarettes smoked
Pharmacist Time | 6 months
  Time spent by pharmacists in counselling patients

CONTACTS AND LOCATIONS:
Overall Officials: Shawn C Bugden, PharmD, Principal Investigator — College of Pharmacy, University of Manitoba
Locations (1):
- College of Pharmacy, University of Manitoba, Winnipeg, Manitoba, Canada